CLINICAL TRIAL: NCT03352700
Title: Premedication Dyclonine Improves Visibility During Bowel Cleansing for Colonoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Director, Head of Department of Gastroenterology, Principal Investigator, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Dyclonine-01
Record Dates: First submitted 2017-11-21; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Bowel Preparation Scale; the Amount of Air Bubble; Adenoma Detection Rate

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3L PEG (Placebo Comparator): only used 3L PEG
  Interventions: Drug: 3L PEG
- 3L PEG+Dyclonine Hydrochloride Mucilage (Experimental): used 3L PEG+Dyclonine Hydrochloride Mucilage
  Interventions: Drug: 3L PEG+Dyclonine Hydrochloride Mucilage

INTERVENTIONS:
Drug: 3L PEG — Group A patients (n = 300) used only 3L PEG before colonoscopy.
  Arms: 3L PEG
Drug: 3L PEG+Dyclonine Hydrochloride Mucilage — Patients in group B (n = 300) were additionally advised to Dyclonine Hydrochloride Mucilage plus 3 L PEG
  Arms: 3L PEG+Dyclonine Hydrochloride Mucilage

SUMMARY:
In this randomized controlled study, consecutive outpatients scheduled for elective colonoscopy were randomized into two groups. Group A patients (n = 300) used only 3L PEG before colonoscopy. Patients in group B (n = 300) were additionally advised to Dyclonine Hydrochloride Mucilage plus 3L PEG, The overall quality of colonoscopy cleaning was evaluated using the Boston Bowel Preparation Scale by a single endoscopist who was blinded to the intervention. Visibility was blindly assessed for the amount of air bubbles and adenoma detection rate (ADR). Difficulty of procedure, and adverse events were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are between 18-75 years old
2. undergoing colonoscopy for diagnostic investigation, colorectal cancer screening or follow-up

Exclusion Criteria:

1. suspected gastrointestinal obstruction or perforation
2. severe acute inflammatory bowel disease
3. toxic megacolon
4. ileus or gastric retention, ileostomy,
5. hypersensitivity to any of the ingredients
6. pregnancy and lactation and/or at a risk of becoming pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
the amount of air bubbles | 2 days
  The amount of intraluminal air bubbles was classified into four grades as shown below: Grade 0 = No or minimal scattered bubbles; Grade 1 = Bubbles covering at least half the luminal diameter; Grade 2 = Bubbles covering the circumference of the lumen; Grade 3 = Bubbles filling the entire lumen. Bubbles filling the entire lumen.

SECONDARY OUTCOMES:
adenoma detection rate | 2 days
  The secondary end point of the study included adenoma detection rate
mean total adenomas detected beyond first | 2 days
  It was a new metric called ADR-Plus, the mean number of incremental adenomas after the fist.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Cheng, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China